CLINICAL TRIAL: NCT03673735
Title: A Randomized Phase III Study on Maintenance Durvalumab vs Placebo Following Post-operative Concomitant Chemoradiation in Subjects With HPV-negative Squamous Cell Head and Neck Carcinoma (HNSCC) With High Risk of Recurrence
Brief Title: Maintenance Immune Check-point Inhibitor Following Post-operative Chemo-radiation in Subjects With HPV-negative HNSCC
Acronym: ADHERE
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Company withdrew interest
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EORTC 1735-HNCG; 2018-002730-21 (EudraCT Number)
Record Dates: First submitted 2018-08-03; First posted 2018-09-17 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Squamous Cell Head and Neck Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — durvalumab; Radiotherapy; Saline Solution; Cisplatin; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Arm (Experimental): Patients will receive 1 infusion of 1500 mg Durvalumab within 1 week prior to concurrent chemoradiotherapy. Chemoradiation should start within 6 weeks after surgery and within 1 week maximum of the induction phase. Radiation will consist of 33 fractions over 6 weeks for a total of 66 Gy. Chemotherapy will consist of cisplatin 100 mg/m2 given on days 1, 22 and 43 of radiotherapy. Maintenance phase with Durvalumab will begin within 1 to 28 days maximum after the end of radiotherapy and will consist of 6 doses administered every 4 weeks.
  Interventions: Drug: Durvalumab; Radiation: radiotherapy; Drug: Cisplatin
- Control arm (Placebo Comparator): Patients will receive 1 infusion of placebo within 1 week prior to concurrent chemoradiotherapy. Chemoradiation should start within 6 weeks after surgery and within 1 week maximum of the induction phase. Radiation will consist of 33 fractions over 6 weeks for a total of 66 Gy. Chemotherapy will consist of cisplatin 100 mg/m2 given on days 1, 22 and 43 of radiotherapy. Maintenance phase with placebo will begin within 1 to 28 days maximum after the end of radiotherapy and will consist of 6 doses administered every 4 weeks.
  Interventions: Radiation: radiotherapy; Drug: Placebo; Drug: Cisplatin

INTERVENTIONS:
Drug: Durvalumab — Durvalumab (one dose) before CRT and for 6 months Q4W after CRT
  Other Names: MEDI4736
  Arms: Experimental Arm
Radiation: radiotherapy — radiotherapy is administered in 33 fractions over 6.5 weeks fro a total of 66 Gy
Drug: Placebo — placebo (one dose) before CRT and for 6 months Q4W after CRT
  Other Names: saline solution
  Arms: Control arm
Drug: Cisplatin — Cisplatin (100mg/m2) is administered at day 1, 22, 43 of radiotherapy
  Other Names: chemotherapy

SUMMARY:
This is a phase III randomized blind placebo-controlled study, designed to show the superiority of the experimental arm to the control arm.

After surgery and checking eligibility criteria, patients will be randomized between the control and the experimental arms with a 1:1 ratio (randomization will take place at a maximum 4 weeks after surgery):

* Experimental Arm: Durvalumab (one dose) before chemoradiotherapy (CRT) and for 6 months every 4 weeks (Q4W) after CRT
* Control Arm: placebo (one dose) before CRT and for 6 months Q4W after CRT Radiotherapy planning will take place after randomization. The primary endpoint of this trial is disease free survival (DFS), measured from the date of randomization to the date of first occurrence of any loco-regional recurrence, metastatic progression, or death due to any cause.

ELIGIBILITY:
Inclusion Criteria:

* Patients with squamous cell carcinoma of the oral cavity (excluding lip), larynx, hypopharynx or p16-negative oropharynx (p16 determined locally)
* Surgical treatment no more than 4 weeks prior randomization (which may include revisions, secondary flaps etc., VACs) with completed wound healing no later than 4 weeks after the initial procedure
* At high risk of locoregional recurrence based on extranodal extension (ENE) and/or R1 resection margin < 1 mm, as documented in the pathology report of surgery.
* With postoperative pathology stage III or IV or stage II but with positive margins (based on AJCC 8th edition)
* Availability of FFPE tumor tissue block from the resection specimen
* Availability of operative and pathology report and preoperative diagnostic images for retrospective review
* ECOG Performance status 0-1
* Age ≥ 18 years
* Adequate bone marrow, liver and renal functions within 7 days from randomization
* Audiogram must be within normal range
* Chemoradiation planned to start within maximum of 2 weeks from randomization. Whenever indicated, dental extraction should be carried out at least 10 days before the start of CRT.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients within 72 hours prior to randomization.
* Patients of childbearing / reproductive potential must agree to use highly effective methods of contraception based on the Clinical trials Facilitation Group (CFTG) guidance from randomization up to 90 days after the last dose of Durvalumab/placebo (Appendix I) or 6 months after the last CRT, whichever is longer.
* Female subjects who are breast feeding should discontinue nursing prior to randomization to 90 days after the last dose of Durvalumab.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with CRT or Durvalumab may be included only after consultation with the clinical research physician
* Before patient randomization, written informed consent must be given according to ICH/GCP, and national/local regulations

Exclusion Criteria:

* Evidence of distant metastases before and after surgery
* Any evidence of early locoregional recurrence after surgery
* Any prior treatment with chemotherapy, radiotherapy or cetuximab
* Any previous treatment with a PD1 or PD-L1 inhibitor, including Durvalumab, a CTLA-4 inhibitor including tremelimumab or other checkpoint inhibitors or other immunotherapy during the last 12 months
* Any contraindication to cisplatin and radiotherapy
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Body weight </=30 kg
* Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Current or prior use of immunosuppressive medication within 14 days prior to enrollment, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid, or steroids as premedication for hypersensitivity reactions (eg, CT scan premedication)
* History of allogenic organ transplantation
* Receipt of live attenuated vaccination within 30 days prior to enrollment Note: Patients, if enrolled, should not receive live vaccine whilst receiving Durvalumab and up to 30 days after the last dose of Durvalumab.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis, systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.). Following disorders are acceptable:
* Vitiligo or alopecia
* Hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement
* Any chronic skin condition that does not require systemic therapy
* Active disease in the last 5 years may be included but only after consultation with the treating physician
* Celiac disease controlled by diet alone
* Diverticulosis
* Known allergy or hypersensitivity to cisplatin and Durvalumab or any of its excipients
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension (defined as blood pressure above 160/90 mm Hg despite medication), unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, active peptic ulcer disease or gastritis, liver cirrhosis CHILD B+, C, active bleeding diatheses
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* History of another primary malignancy with the exception of:
* Malignancy treated with curative intent and with no known active disease ≥5 years before enrollment and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease
* History of symptomatic brain metastases and leptomeningeal carcinomatosis
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Female subjects who are pregnant or male or female subjects of reproductive potential who are not willing to employ effective birth control from randomisation to 90 days after the last dose of Durvalumab
* Any psychological, familial, sociological or geographical condition that could increase risk of incurring AEs or compromise the ability of the patient to give written informed consent, or hamper compliance with the study protocol and follow-up schedule; these conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
disease free survival | 3 years and half after last pateint in
  The main study objective is to test whether treatment with Durvalumab, given before and after completion of standard adjuvant chemoradiation, significantly prolongs disease free survival in macroscopically completely resected HPV negative advanced head and neck cancer at high risk of recurrence.

SECONDARY OUTCOMES:
overall survival | 5 years after last patients in
  To assess the impact of postoperative Durvalumab on the overall survival
Cumulative incidence of distant metastases | 5 years after last patients in
  Time to distant metastases is defined as the time interval between the date of randomization and the first date when distant disease is detected. Cumulative incidence of distant metastases is estimated considering death or diagnosis of loco-regional recurrence in absence of distant disease is considered as a competing risk event. If a recurrence is detected at the same time at both loco-regional and distant sites, this is considered as a competing risk for this endpoint.
Cumulative incidence of loco-regional recurrence | 5 years after last patients in
  Time to loco-regional recurrence is the time interval between the date of randomization and the date where local or regional recurrence is first detected. Cumulative incidence of loco-regional recurrence is estimated considering death or diagnosis of distant metastases in absence of loca l or regional recurrence is considered as a competing risk event. If a recurrence is detected at the same time at both loco-regional and distant sites, this is considered as an event of interest for this endpoint.
Cumulative incidence of second cancers (all sites) | 5 years after last patients in
  first diagnosis of any second cancer in the head and neck region or outside the head and neck region. Cumulative incidence of second cancer is estimated considering death without a second cancer is considered as a competing risk.
Rate of toxicity assessed by clinicians | 5 years after last patients in
  All adverse events will be recorded; the investigator will assess whether those events are drug related (reasonable possibility, no reasonable possibility) and this assessment will be recorded in the database for all adverse events. Adverse events will be recorded according to NCI-CTCAE
Health-related quality of Life questionnaires: QLQ-C30 | 5 years after last patients in
  To compare the addition of immunotherapy to chemo-radiation therapy on health-related quality of life. Quality of life will be assessed with the EORTC Quality of Life Questionnaire (QLQ-C30) version 3.
  The EORTC Quality of Life Questionnaire (QLQ-C30) version 3 is patient questionnaire composed of 30 single questions which form 15 multi-item and single-item scales. These include five functional scales (physical, role, emotional, social, and cognitive), three multi-item symptom scales (fatigue, nausea and vomiting and pain), six single item symptom scales (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties) and a global health status/QoL scale. The scoring algorithm for the scales results in a score from 0 to 100 where a high score for a functional scale represents a healthy level of functioning, but a high score for a symptom scale represents a high level of problems.

IPD SHARING:
Plan to Share IPD: No